CLINICAL TRIAL: NCT06221488
Title: THWART-TB: Testing Health Workers At Risk to Advance Our Understanding of TB Infection
Brief Title: Testing Health Workers At Risk to Advance Our Understanding of TB Infection
Acronym: THWART-TB
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Ruvandhi Nathavitharana, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: DP2AI176896 (NIH)
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis; Tuberculosis Infection
Keywords: Tuberculosis; TB; TB infection; Health worker
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will collect blood (whole blood, plasma, serum, PBMCs), sputum, and nasopharyngeal swab specimens. Specimens will be stored for future use, which will remain in South Africa for future research and training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health workers: Health workers with baseline negative interferon gamma release assays
  Interventions: Diagnostic Test: TB infection testing

INTERVENTIONS:
Diagnostic Test: TB infection testing — Diagnostic testing with existing and novel tests to evaluate for TB infection and disease

SUMMARY:
It has been estimated that 1.7 billion people have tuberculosis (TB) infection; yet current tests are unable to predict which people are at highest risk of developing TB disease, which can be life-threatening. THWART-TB is a prospective longitudinal cohort study of health workers (HWs) in Cape Town, South Africa, where our preliminary data reveals HWs have a high annual TB infection risk (34%). This cohort, who will undergo frequent serial evaluation (every 3 months) with a combination of novel assays never previously evaluated together, presents a unique opportunity to evaluate immune responses at the time of initial infection and to characterize the dynamic profile of these immune responses over time in a high-risk population. The knowledge generated will improve our understanding of TB infection and help to identify which people exposed to TB may remain at risk, enabling us to better target preventive strategies.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a leading infectious cause of death in South Africa and globally.1.7 billion people worldwide are estimated to have been infected with TB (LTBI). However, current LTBI tests cannot distinguish between current infection versus a persistent immune response to a cleared infection and have a low predictive value to identify which people are at future risk of developing active TB disease. Moreover, LTBI following exposure to Mycobacterium tuberculosis (Mtb) is not a steady state process. The dynamic host-pathogen interactions that lead to bacterial clearance, suppression, or disease are not understood. The investigators propose to establish a prospective longitudinal cohort study of health workers (HWs) in Cape Town, South Africa, where previous data demonstrated HWs have a high annual TB infection risk (34%). Our fundamentally innovative approach will characterize early TB infection using serial testing every 3 months for one year with a combination of established and novel assays never previously evaluated together. This presents a unique opportunity to evaluate host and pathogen responses at the time of initial infection and to characterize the dynamic profile of these responses over time in a high-risk population, establishing a longitudinal platform for future studies, including through biobanked specimens. This study will generate critical data of local relevance given the devastating ongoing impact of TB in South Africa.

The investigators hypothesize that Mtb persistence or clearance in the first year after incident infection (determined by follow up interferon gamma release assay (IGRA) after a new IGRA conversion) correlates with dynamic changes in host blood transcriptional markers of incipient and active TB, Mtb antibody responses and Mtb DNA detection.

Aim 1: To evaluate the temporal dynamics of established and novel interferon-gamma based tests for latent TB infection. The investigators hypothesize high-frequency serial IGRA testing will enable us to identify how often sustained conversions and reversions occur after early TB infection (based on initial IGRA conversion) over 1 year follow up. The investigators will compare the performance of established and novel IGRAs and new LTBI tests.

Aim 2: To evaluate the temporal dynamics of host responses to TB based on RNA biosignatures and Mtb antibodies. The investigators hypothesize that sustained IGRA conversion may predict seroconversion and a contemporary rise in host-response blood transcriptional biomarkers of TB and will evaluate how these profiles change over time

Aim 3: To evaluate the temporal dynamics of novel assays to detect pathogen-directed Mtb DNA markers of early infection. The investigators hypothesize IGRA conversion, seroconversion, or rise in host-response blood transcriptional biomarkers of TB will predict detection of Mtb DNA using a range of novel assays to identify a pathogen-derived marker of early infection that is complementary to evaluation of the host immune response.

The investigators will conduct a prospective cohort study recruiting HWs at Tygerberg Hospital in Cape Town, where our prior study demonstrated the feasibility of recruiting this population. The investigators will recruit equal numbers of men and women and ensure participant diversity reflective of the South African population. The investigators will conduct serial testing every 3 months (based on a systematic review suggesting this testing interval may be optimal while being pragmatically feasible) with a combination of established and novel assays chosen to evaluate host and pathogen-derived signatures never evaluated before in parallel to identify correlates of risk and protection: IGRAs, novel LTBI tests, blood RNA biosignatures, Mtb-specific antibody responses and Mtb DNA detection assays. HWs are a unique population to understand serial host and pathogen dynamics including whether tests revert to negative i.e. whether initial IGRA conversions are transient versus persistent, and whether re-conversions may potentially represent reinfection given high exposure risk.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Health worker
* Able to provide informed consent

Exclusion Criteria:

* Prior history of TB or known prior positive IGRA
* Current or prior history of taking anti-TB treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be health workers (primarily clinical but may include support staff) who are >18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Interferon gamma release assay conversion | Tested at months 0, 3, 6, 9, 12, 24
  IGRA conversion using Quantiferon-Plus

SECONDARY OUTCOMES:
TB disease | Assessed at months 0, 3, 6, 9, 12, 24
  Development of active TB disease, defined by positive Xpert Ultra or defined clinically based on clinician starting treatment for active TB disease with combination of suggestive symptoms and/or abnormalities on chest x-ray in the absence of bacteriological confirmation.

CONTACTS AND LOCATIONS:
Overall Officials: Ruvandhi Nathavitharana, MBBS MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Stellenbosch University, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nathavitharana RR, Mishra H, Sullivan A, Hurwitz S, Lederer P, Meintjes J, Nardell E, Theron G. Predicting Airborne Infection Risk: Association Between Personal Ambient Carbon Dioxide Level Monitoring and Incidence of Tuberculosis Infection in South African Health Workers. Clin Infect Dis. 2022 Oct 12;75(8):1297-1306. doi: 10.1093/cid/ciac183. PMID 35348657